CLINICAL TRIAL: NCT00689793
Title: Clinical Evaluation of Iron Treatment Efficiency Among Non-anemic But Iron-deficient Female Blood Donors : a Randomized Controlled Trial
Brief Title: Clinical Evaluation of Iron Treatment Efficiency Among Non-anemic But Iron-deficient Female Blood Donors
Acronym: ferdon
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: Pierre Fabre Laboratories (Industry)
Responsible Party: Principal Investigator, Bernard Favrat, MD, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Iron-0508-PMU
Record Dates: First submitted 2008-05-28; First posted 2008-06-04 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-01

CONDITIONS: Fatigue; Iron Deficiency
Keywords: Fatigue; Blood donation; Iron deficiency; Ferrous sulphate; Donation; Donors; Iron; Ferritin; Hemoglobin; Anemia; Anaemia; Haemoglobin; Don; Women blood donors
MeSH Terms: conditions — Fatigue; Iron Deficiencies; Anemia | interventions — ferrous sulfate; ferrous sulfate, mucin drug combination; Iron, Dietary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Ferrous sulphate
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferrous sulphate — Volunteers will receive 80 mg/day oral ferrous sulphate (Tardyferon®) for four weeks. Visual analogical scales and questionnaires will be performed at day 0 and 30 to quantify fatigue (" Fatigue Severity Scale"). We will also check depression and anxiety symptoms (" Prime MD ") and health survey (" SF-12 "). An evaluation of the menstruation (" Pictorial Bleeding Assessment Chart " of Jansen) will be performed at day 0 to detect a possible hypermenorrhea (appendix 1-4). A physical test will be performed (Chester Step Test) to assess the VO2 max. Every side effect will be written on follow-up notes.
  Other Names: Iron treatment; Ferrous sulphate treatment; Tardyferon; Robapharm; Fer; Sulphate de fer; Sulphate ferreux; Iron deficiency
  Arms: 1
Drug: Placebo — Volunteers will receive 1 pill/day oral placebo for four weeks. Visual analogical scales and questionnaires will be performed at day 0 and 30 to quantify fatigue (" Fatigue Severity Scale"). We will also check depression and anxiety symptoms (" Prime MD ") and health survey (" SF-12 "). An evaluation of the menstruation (" Pictorial Bleeding Assessment Chart " of Jansen) will be performed at day 0 to detect a possible hypermenorrhea (appendix 1-4). A physical test will be performed (Chester Step Test) to assess the VO2 max. Every side effect will be written on follow-up notes.
  Other Names: Iron treatment; Ferrous sulphate treatment; Tardyferon; Robapharm; Fer; Sulphate de fer; Sulphate ferreux; Iron deficiency
  Arms: 2

SUMMARY:
The purpose of this study is to determine the subjective response of iron substitution (Tardyferon®) on fatigue in women blood donors with a mean serum ferritin < 30ng/ml and to assess variation of ferritin and hemoglobin after a blood donation.

DETAILED DESCRIPTION:
* Actually, there's no recommendation to check ferritin level in blood donors, even if several studies pointed out the high prevalence of iron deficiency after a blood donation. Furthermore, some clinical trials showed that non-anaemic women with unexplained fatigue may benefit from iron supplementation.
* The purpose of this study is to determine the subjective response of iron substitution (Tardyferon®) on fatigue in women blood donors with a mean serum ferritin < 30ng/ml and to assess variation of ferritin and hemoglobin after a blood donation.
* We will measure blood count, ferritin level and C-reactive protein at the time of the blood donation and then after a week, a month and 3 months.

A week after the blood donation, donors with a ferritin level <30 ng/ml and hemoglobin > 120g/l (non anaemic) will be included in the study and randomised. A one-month iron treatment vs placebo will be introduced. To assess the subjective response on fatigue, the donors will fill in different questionnaires at the time of the blood donation and then after a week, a month and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* women
* aged 18 - 50
* eligible for a blood donation

Exclusion Criteria:

* men
* age below 18 or above 50
* not eligible for a blood donation (according to the blood donation eligibility guidelines of the Swiss Red Cross)
* hemochromatosis, psychiatric / thyroid / hepatic / rheumatismal / kidney or cardiopulmonary diseases that can cause fatigue
* intestinal disease or medical treatment that can perturb iron absorption and/or excretion
* donors with mental disorder or psychiatric disease that are unable to give consent
* acute or chronic inflammation
* diabetes and pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Favrat, MD PD, Principal Investigator — Department of Amulatory Care and Community Medicine, University of Lausanne; Baptiste Pedrazzini, MD, Study Chair — Department of Amulatory Care and Community Medicine, University of Lausanne; Jacques Cornuz, Prof, Study Chair — Department of Amulatory Care and Community Medicine, University of Lausanne; Alain Pécoud, Prof, Study Chair — Department of Amulatory Care and Community Medicine, University of Lausanne; Sophie Waldvogel, MD, Study Chair — Blood Transfusion Department, University Hospitals of Lausanne; Jean-Daniel Tissot, Prof, Study Chair — Blood Transfusion Department, University Hospitals of Lausanne
Locations (1):
- Department of Ambulatory Care and Community Medicine, University Hospitals of Lausanne, Lausanne, Bugnon 44, Switzerland

REFERENCES:
- [Background] Verdon F, Burnand B, Stubi CL, Bonard C, Graff M, Michaud A, Bischoff T, de Vevey M, Studer JP, Herzig L, Chapuis C, Tissot J, Pecoud A, Favrat B. Iron supplementation for unexplained fatigue in non-anaemic women: double blind randomised placebo controlled trial. BMJ. 2003 May 24;326(7399):1124. doi: 10.1136/bmj.326.7399.1124. PMID 12763985
- [Background] Patterson AJ, Brown WJ, Powers JR, Roberts DC. Iron deficiency, general health and fatigue: results from the Australian Longitudinal Study on Women's Health. Qual Life Res. 2000;9(5):491-7. doi: 10.1023/a:1008978114650. PMID 11190004
- [Background] BEUTLER E, LARSH SE, GURNEY CW. Iron therapy in chronically fatigued, nonanemic women: a double-blind study. Ann Intern Med. 1960 Feb;52:378-94. doi: 10.7326/0003-4819-52-2-378. No abstract available. PMID 13800263
- [Background] Bruner AB, Joffe A, Duggan AK, Casella JF, Brandt J. Randomised study of cognitive effects of iron supplementation in non-anaemic iron-deficient adolescent girls. Lancet. 1996 Oct 12;348(9033):992-6. doi: 10.1016/S0140-6736(96)02341-0. PMID 8855856
- [Background] Patterson AJ, Brown WJ, Roberts DC. Dietary and supplement treatment of iron deficiency results in improvements in general health and fatigue in Australian women of childbearing age. J Am Coll Nutr. 2001 Aug;20(4):337-42. doi: 10.1080/07315724.2001.10719054. PMID 11506061
- [Background] Newman BH, Roth AJ. Estimating the probability of a blood donation adverse event based on 1000 interviewed whole-blood donors. Transfusion. 2005 Nov;45(11):1715-21. doi: 10.1111/j.1537-2995.2005.00595.x. PMID 16271095
- [Background] Newman B. Iron depletion by whole-blood donation harms menstruating females: the current whole-blood-collection paradigm needs to be changed. Transfusion. 2006 Oct;46(10):1667-81. doi: 10.1111/j.1537-2995.2006.00969.x. No abstract available. PMID 17002622
- [Background] Maghsudlu M, Nasizadeh S, Toogeh GR, Zandieh T, Parandoush S, Rezayani M. Short-term ferrous sulfate supplementation in female blood donors. Transfusion. 2008 Jun;48(6):1192-7. doi: 10.1111/j.1537-2995.2007.01671.x. Epub 2008 Mar 17. PMID 18363581
- [Background] Magnussen K, Bork N, Asmussen L. The effect of a standardized protocol for iron supplementation to blood donors low in hemoglobin concentration. Transfusion. 2008 Apr;48(4):749-54. doi: 10.1111/j.1537-2995.2007.01601.x. Epub 2008 Jan 8. PMID 18194390
- [Background] Brownlie T 4th, Utermohlen V, Hinton PS, Giordano C, Haas JD. Marginal iron deficiency without anemia impairs aerobic adaptation among previously untrained women. Am J Clin Nutr. 2002 Apr;75(4):734-42. doi: 10.1093/ajcn/75.4.734. PMID 11916761
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Background] Janssen CA. A simple visual assessment technique to discriminate between menorrhagia and normal menstrual blood loss. Eur J Obstet Gynecol Reprod Biol. 1996 Dec;70(1):21-2. doi: 10.1016/s0301-2115(96)02570-5. No abstract available. PMID 9031914
- [Background] Buckley JP, Sim J, Eston RG, Hession R, Fox R. Reliability and validity of measures taken during the Chester step test to predict aerobic power and to prescribe aerobic exercise. Br J Sports Med. 2004 Apr;38(2):197-205. doi: 10.1136/bjsm.2003.005389. PMID 15039259
- [Result] Waldvogel S, Pedrazzini B, Vaucher P, Bize R, Cornuz J, Tissot JD, Favrat B. Clinical evaluation of iron treatment efficiency among non-anemic but iron-deficient female blood donors: a randomized controlled trial. BMC Med. 2012 Jan 24;10:8. doi: 10.1186/1741-7015-10-8. PMID 22272750
- [Derived] Pedrazzini B, Waldvogel S, Cornuz J, Vaucher P, Bize R, Tissot JD, Pecoud A, Favrat B. The impact of iron supplementation efficiency in female blood donors with a decreased ferritin level and no anaemia. Rationale and design of a randomised controlled trial: a study protocol. Trials. 2009 Jan 16;10:4. doi: 10.1186/1745-6215-10-4. PMID 19149890

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Premopausal female blood donors coming spontaneously to the donation center, were asked to participated to this study. After agreement an informed consent was signed.
Pre-assignment Details: One week after whole blood donation, participants were randomized if they were not anemic and their ferritin level was < or = 30 ng/mL.
Groups:
- Oral Treatment of Iron: One week after donation, donors self-administered ferrous sulfate (80mg of elemental iron daily) during one month.
- Placebo: One week after donation, donors self-administered on pill of placebo (daily), during one month.
Period: Overall Study
Arm/Group | Oral Treatment of Iron | Placebo
Started | 78 | 76
Completed | 74 | 71
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Treatment of Iron | Placebo | Total
Number analyzed (Participants) | 78 | 76 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 76 | 154
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.9 (8.4) | 30.7 (8.8) | 31.6 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 76 | 154
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 78 | 76 | 154

OUTCOME MEASURES:

1. Primary Outcome: Level of Fatigue Before and After Iron Treatment/Placebo, Using a 10 Point Visual Analogue Scale.
Description: The level of fatigue perceived at baseline and after 4 weeks was scored on a 10-point visual analogue scale ranging from "no fatigue=0" to "very severe fatigue=10".
Time Frame: baseline and 4 weeks
Population: The sample size for randomized volunteers was calculated using a two-sample comparison of means to detect a one point difference in the visual analogical scale (first outcome).
Measure: Mean (Standard Deviation); unit: centimeter
Groups:
- Placebo: One week after donation, donors self-administered one pill of placebo (daily), during 4 weeks.
Arm/Group | Oral Treatment of Iron | Placebo
Number analyzed (Participants) | 74 | 71
centimeter | 3.4 (2.4) | 3.5 (2.5)
Statistical Analysis 1: Comparison: Oral Treatment of Iron; The null hypothesis was that there was no difference in fatigue VAS scores between the treatment and placebo groups at 4 weeks; Test type: Superiority or Other; p = 0.69, Regression, Linear — Significant level of treatment effect was set at p<0.05; Level of fatigue at four weeks:dependant variable. Group allocation and level of fatigue at baseline: independant variables; Mean Difference (Final Values) = 1, 95% CI 2-sided [0 to 10], Standard Deviation 2.5

2. Secondary Outcome: Hemoglobin Variation Before and After Treatment vs Placebo
Description: The level of hemoglobin measured 4 weeks after randomization
Time Frame: baseline and 4 weeks
Population: The number of participants was calculated according to the primary outcome.
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- Oral Treatment of Iron: One week after donation, donors self-administered ferrous sulfate (80mg of elemental iron daily), during one month.
Arm/Group | Oral Treatment of Iron | Placebo
Number analyzed (Participants) | 74 | 71
g/L | 135 (6.7) | 130 (5.3)
Statistical Analysis 1: Comparison: Oral Treatment of Iron vs Placebo; Test type: Superiority or Other; p < 0.05, Regression, Linear; Hemoglobin value at four weeks : dependant variable. Group allocation and hemoglobin value at baseline : independant variables; Mean Difference (Final Values) = 3, 95% CI [0 to 10], Standard Deviation 6.5

3. Secondary Outcome: Ferritin Change Before and After 4 Weeks of Treatment/Placebo
Description: Level of ferritin measured 4 weeks after randomization
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oral Treatment of Iron | Placebo
Number analyzed (Participants) | 74 | 71
ng/mL | 28.0 (9.8) | 12.9 (8.3)
Statistical Analysis 1: Comparison: Oral Treatment of Iron vs Placebo; Test type: Superiority or Other; p < 0.05, Regression, Linear; Ferritin level at 4 weeks : dependant variable. Group allocation and ferritin level at baseline: independant variables; Mean Difference (Final Values) = 15, 95% CI 2-sided [0 to 30], Standard Deviation 8

4. Secondary Outcome: Aerobic Capacity Using an Indirect Measurement of VO2Max : Chester Step Test
Description: Subjects were asked to step on to and off a 20cm step at a rate set by a metronome. Step rate increased gradually until subject reached her submaximal predicted heart rate.
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: mLO2/kg/min
Arm/Group | Oral Treatment of Iron | Placebo
Number analyzed (Participants) | 74 | 71
mLO2/kg/min | 40.5 (14.5) | 40.1 (17)
Statistical Analysis 1: Comparison: Oral Treatment of Iron vs Placebo; Test type: Superiority or Other; p = 0.05, Regression, Linear; Aerobic capacity at 4 weeks : dependant variables. Group allocation and aerobic capacity at baseline : independant variable; Mean Difference (Final Values) = 3, 95% CI 2-sided [0 to 6], Standard Deviation 3

5. Secondary Outcome: Response of Iron Supplementation on Mental Disorder
Description: Depression was assessed using the Prime-MD Patient Health Questionnaire (PHQ-9), self-administered by the subject.Diagnosis of depression syndrom was made scoring results of the nine item (range : 0-3). A score >15 (range of total overall scale:0-27) was considered as a depression syndrome. The outcome measure is the number the donors with a depression syndrome at baseline who had a positive response (total score= or <15) after placebo or treatment.
Time Frame: baseline and 4 weeks
Population: Number of participant was set according the primary outcome.
Measure: Number; unit: participants
Arm/Group | Oral Treatment of Iron | Placebo
Number analyzed (Participants) | 74 | 71
participants | 3 | 4

6. Secondary Outcome: Adherence to Treatment.
Description: Adherence to treatment was calculated as the number of days with at least one opening of the electronic device divided by the total number of monitored days. The device was a MEMS (Medication Event Monitoring System,AARDEX, Europe, Switzerland)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of day
Arm/Group | Oral Treatment of Iron | Placebo
Number analyzed (Participants) | 74 | 71
percentage of day | 96 (16.7) | 96 (14.2)

ADVERSE EVENTS:
Time Frame: adverse events were reported during the 4 weeks of treatment/placebo
Arm/Group | Oral Treatment of Iron | Placebo
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/71
Other Adverse Events (participants affected / at risk) | 29/74 | 11/71
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Treatment of Iron (N=74) | Placebo (N=71)
gastro-intestinal events (Gastrointestinal disorders) | 25 (25) | 11 (11)
other events (not serious) (General disorders) | 6 (6) | 3 (3) — dizziness (n=3), headache (n=2), acne (n=2), palpitations (n=1), and renal lithiasis (n=1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No